CLINICAL TRIAL: NCT02148679
Title: Effects of Home-delivered Low-sodium Meals in Older Adults Following Heart Failure Hospitalization.
Brief Title: Geriatric Out of Hospital Randomized Meal Trial in Heart Failure
Acronym: GOURMET-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: PurFoods, LLC (Unknown); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Scott L. Hummel, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HUM00083272; R21AG047939 (NIH)
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Heart Failure
Keywords: Heart Failure; Diet
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- DASH/SRD (Experimental): Patients receive Heart Failure Society of America pamphlet, "How to eat a low sodium diet" at hospital discharge
  Study staff will phone patients at weeks 2 and 3 to confirm patients' understanding of dietary instructions
  Intervention: pre-prepared, home delivered DASH/SRD-compliant meals for 4 weeks after hospital discharge
  Interventions: Other: DASH/SRD
- Attention Control (Placebo Comparator): Patients receive Heart Failure Society of America pamphlet, "How to eat a low sodium diet" at hospital discharge
  Study staff will phone patients at weeks 2 and 3 to confirm patients' understanding of dietary instructions
  Interventions: Other: DASH/SRD; Other: Usual care

INTERVENTIONS:
Other: DASH/SRD — Study food for this investigation will be designed and prepared by PurFoods, LLC (Des Moines, IA) dietitians under the direction of Dr. Sam Beattie, Ph. D., and in consultation with research dietitians at the University of Michigan and Columbia University. Study patients randomized to food delivery will select from an available menu of meal options that adhere to nutritional targets as above. Study food will be pre-packaged for storage with preparation (typically microwave heating) to be completed at home by the subject, and will be delivered every 1 to 2 weeks under the direction of PurFoods.
  Other Names: Mom's Meals
Other: Usual care — Standardized advice to restrict dietary sodium intake to < 2000 mg/day
  Arms: Attention Control

SUMMARY:
Study subjects will receive either pre-prepared, home-delivered DASH/SRD-compliant meals or attention control for 4 weeks after hospital discharge.

DETAILED DESCRIPTION:
This is a three center, randomized, single-blind, attention controlled trial of 12 weeks total duration designed to determine the safety and efficacy of home-delivered sodium-restricted Dietary Approaches to Stop Hypertension (DASH/SRD)-compliant meals in older adults (age >= 65 years) following discharge from a hospital admission for acutely decompensated heart failure. 66 subjects will be randomized in a 1:1 stratified fashion by gender and left ventricular ejection fraction (< vs. ≥ 50%).

107 subjects yielded 66 randomized subjects.

Study subjects will receive either pre-prepared, home-delivered DASH/SRD-compliant meals or attention control for 4 weeks after hospital discharge. The three study sites will be Columbia University Medical Center, the Ann Arbor Veterans Affairs Health System, and the University of Michigan Health System. Investigators will be blinded to group assignment, food diaries, and urinary electrolyte measurements until the completion of the study

ELIGIBILITY:
Inclusion Criteria:

66 male and female patients aged ≥ 55 years with history of systemic hypertension and acutely decompensated heart failure (ADHF; primary diagnosis for admission or secondary diagnosis after hospitalization for another reason). ADHF will be confirmed by the study physician and defined as a combination of symptoms, signs, and HF-specific medical treatments. Specifically, ADHF will require that all four of the following conditions are met:

* ≥1 symptom of HF (dyspnea, fatigue, orthopnea, paroxysmal nocturnal dyspnea) has worsened from baseline
* ≥ 2 signs of HF (pulmonary congestion on exam and/or chest X-ray, elevated jugular venous pressure, peripheral edema or rapid weight gain, and/or increased B-type natriuretic peptide (BNP; ≥100 pg/ml)
* change in medical treatment specifically targeting HF (diuretics, vasodilators, and/or neurohormonal modulating agents)
* no other cause of the patient's symptoms and signs is apparent

Exclusion Criteria:

* persistent hypotension during hospitalization or excessive risk of hypotension from the study diet as judged by the investigators or systolic BP <110 on discharge
* use of inotropic therapy at hospital discharge,
* severe valvular heart disease as the primary etiology of the patient's HF syndrome
* uncontrolled hypertension defined as the following criteria for the last 24 hours prior to discharge (systolic BP >180 mmHg or diastolic BP >100 mmHg)
* having two or more results of a serum potassium >5.0 mmol/L during hospitalization or history of serum potassium >6.0 mmol/L, and/or at an excessive risk of hyperkalemia as judged by the investigators
* severe renal insufficiency (estimated glomerular filtration rate <30 ml/min/1.73m^2 at discharge)
* severe anemia (hemoglobin < 9 gm/dl)
* length of stay <48 hours or >14 days
* co-morbidity with expected survival < 12 months
* active alcohol or substance abuse
* history of persistent noncompliance with treatment recommendations as judged by the investigators

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — eligibility is based on self-representation of gender identity.
Enrollment: 107 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-05-21 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
change in the Kansas City Cardiomyopathy Questionnaire (KCCQ) summary scores for health-related QOL in patients with chronic HF | from study enrollment to 4 weeks post-discharge
  The KCCQ, a self-administered 23-item instrument, assesses physical limitations, symptoms, self-efficacy, social interference, and overall QOL in HF patients. The KCCQ summary score ranges from 0-100, with higher scores indicating better QOL. The KCCQ summary score independently predicts clinical outcomes such as hospitalization and mortality in outpatients with HF, including those recently hospitalized for acute decompensation. It is a reliable and valid measure in HF patients that is more sensitive to change than other measures of QOL, and is especially responsive in patients with multiple comorbidities. A change in KCCQ score of 5 points is clinically significant and correlates with changes in clinical status, physical function, and outcomes.

SECONDARY OUTCOMES:
Safety Monitoring | Baseline and 1 week post discharge
  Renal function and electrolytes will be assessed at baseline and 1 week post-discharge during a safety visit, in which vital signs and targeted physical examination for volume status will allow adjustment of diuretics as clinically indicated. The dietary intervention will be stopped in any patient who develops new or worsened renal impairment as defined by estimated glomerular filtration rate decrease of ≥50%, hyperkalemia (K >5.7 mmol/L), syncope, or other serious adverse event deemed by the investigators to be related to study participation (note participants are inherently at high risk for rehospitalization or mortality, ~20-25% over the 4-week intervention period of the study, ~30-35% over the total 12-week term of the study). Patients randomized to food delivery will have study food intake suspended if hospitalized and resumed at discharge if no safety concerns as defined above.
Dietary Endpoints | baseline, 4 weeks
  Dietary endpoints will include DASH/SRD adherence as measured by 3-day food diary and urinary electrolyte measures (24-hour urinary sodium and potassium). Food frequency questionnaire to establish baseline dietary intake will be obtained at baseline and 12 weeks.
Mechanism-related endpoints | Baseline to 4 weeks
  Mechanism-related endpoints will include changes from baseline to 4 weeks in clinic and 24-hour blood pressure, noninvasive measures of ventricular function and ventricular-arterial coupling, blood/urine measures of neurohormonal activation, oxidative stress, and systemic inflammation, blood volume measurements (subset n=20), and peripheral blood mononuclear cell (PBMC) RNA profiling (subset n=20)

CONTACTS AND LOCATIONS:
Overall Officials: Scott L Hummel, MD, MS, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - Ann Arbor Veterans Affairs Health System, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Columbia University, New York, New York

REFERENCES:
- [Background] Hummel SL, DeFranco AC, Skorcz S, Montoye CK, Koelling TM. Recommendation of low-salt diet and short-term outcomes in heart failure with preserved systolic function. Am J Med. 2009 Nov;122(11):1029-36. doi: 10.1016/j.amjmed.2009.04.025. PMID 19854331
- [Background] Hummel SL, Seymour EM, Brook RD, Kolias TJ, Sheth SS, Rosenblum HR, Wells JM, Weder AB. Low-sodium dietary approaches to stop hypertension diet reduces blood pressure, arterial stiffness, and oxidative stress in hypertensive heart failure with preserved ejection fraction. Hypertension. 2012 Nov;60(5):1200-6. doi: 10.1161/HYPERTENSIONAHA.112.202705. Epub 2012 Oct 1. PMID 23033371
- [Background] Hummel SL, Seymour EM, Brook RD, Sheth SS, Ghosh E, Zhu S, Weder AB, Kovacs SJ, Kolias TJ. Low-sodium DASH diet improves diastolic function and ventricular-arterial coupling in hypertensive heart failure with preserved ejection fraction. Circ Heart Fail. 2013 Nov;6(6):1165-71. doi: 10.1161/CIRCHEARTFAILURE.113.000481. Epub 2013 Aug 28. PMID 23985432
- [Background] Bray GA, Vollmer WM, Sacks FM, Obarzanek E, Svetkey LP, Appel LJ; DASH Collaborative Research Group. A further subgroup analysis of the effects of the DASH diet and three dietary sodium levels on blood pressure: results of the DASH-Sodium Trial. Am J Cardiol. 2004 Jul 15;94(2):222-7. doi: 10.1016/j.amjcard.2004.03.070. PMID 15246908
- [Background] Troyer JL, Racine EF, Ngugi GW, McAuley WJ. The effect of home-delivered Dietary Approach to Stop Hypertension (DASH) meals on the diets of older adults with cardiovascular disease. Am J Clin Nutr. 2010 May;91(5):1204-12. doi: 10.3945/ajcn.2009.28780. Epub 2010 Mar 3. PMID 20200258
- [Background] Racine EF, Lyerly J, Troyer JL, Warren-Findlow J, McAuley WJ. The influence of home-delivered dietary approaches to stop hypertension meals on body mass index, energy intake, and percent of energy needs consumed among older adults with hypertension and/or hyperlipidemia. J Acad Nutr Diet. 2012 Nov;112(11):1755-62. doi: 10.1016/j.jand.2012.06.358. PMID 23102175
- [Background] Wessler JD, Maurer MS, Hummel SL. Evaluating the safety and efficacy of sodium-restricted/Dietary Approaches to Stop Hypertension diet after acute decompensated heart failure hospitalization: design and rationale for the Geriatric OUt of hospital Randomized MEal Trial in Heart Failure (GOURMET-HF). Am Heart J. 2015 Mar;169(3):342-348.e4. doi: 10.1016/j.ahj.2014.11.021. Epub 2015 Jan 7. PMID 25728723
- [Derived] Bilgen F, Chen P, Poggi A, Wells J, Trumble E, Helmke S, Teruya S, Catalan T, Rosenblum HR, Cornellier ML, Karmally W, Maurer MS, Hummel SL. Insufficient Calorie Intake Worsens Post-Discharge Quality of Life and Increases Readmission Burden in Heart Failure. JACC Heart Fail. 2020 Sep;8(9):756-764. doi: 10.1016/j.jchf.2020.04.004. Epub 2020 Jul 8. PMID 32653445
- [Derived] Hummel SL, Karmally W, Gillespie BW, Helmke S, Teruya S, Wells J, Trumble E, Jimenez O, Marolt C, Wessler JD, Cornellier ML, Maurer MS. Home-Delivered Meals Postdischarge From Heart Failure Hospitalization. Circ Heart Fail. 2018 Aug;11(8):e004886. doi: 10.1161/CIRCHEARTFAILURE.117.004886. PMID 30354562